CLINICAL TRIAL: NCT06276868
Title: A Clinical Study of Darsilide Combined With AI, Trastuzumab and Patuzumab in the Neoadjuvant Treatment of HR Positive HER2 Positive Breast Cancer
Brief Title: Darsilide Combined With AI, Trastuzumab and Patuzumab in the Neoadjuvant Treatment of HR+/HER2+ Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-017
Record Dates: First submitted 2023-11-14; First posted 2024-02-26 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
Keywords: HER2-positive Breast Cancer; pathologic complete response; Dalcelli; objective response rate; Disease-free survival
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Intervention Model Description: Prospective, single arm clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalcilib+letrozole+HP (Experimental): All subjects received Dalcilib 150mg qd, stopped for 1 week after 3 weeks，and letrozole (2.5mg qd) (premenopausal combined with OFS). The subjects received 2 cycles of preoperative treatment with darcilib combined with letrozole, trastuzumab, and patstuzumab.
  Then, MRI efficacy evaluation will be conducted, and patients who achieved PR continue to receive the original treatment regimen for 6 cycles, while those who did not achieve PR switched to the TCHP chemotherapy regimen for 6 cycles.
  Interventions: Drug: Dalcilib+letrozole+HP treatment group

INTERVENTIONS:
Drug: Dalcilib+letrozole+HP treatment group — All participants received 150mg of darcilib once a day. Take it continuously for 21 days, then stop taking it for 7 days, with a treatment cycle of 28 days.
  Letrozole 2.5mg once daily (premenopausal patients treated with OFS); Trastuzumab (8mg/kg first dose, 6mg/kg sequential) and Patuzumab (840mg first dose, 420mg/kg sequential) were administered intravenously every 3 weeks, or fixed-dose combination of pertuzumab and trastuzumab for subcutaneous injection (1200 mg pertuzumab plus 600 mg trastuzumab loading dose in 15 mL, followed by 600 mg pertuzumab plus 600 mg trastuzumab maintenance doses in 10 mL), both administered every 3 weeks.
  Other Names: experimental group

SUMMARY:
This study is intended to carry out a single arm, prospective, open clinical study, and use Darsilide combined with endocrine therapy, Trastuzumab and Patuzumab to treat early or locally advanced breast cancer of TPBC before surgery. It is intended to further explore the efficacy and safety of the new adjuvant treatment for TPBC patients with step-down therapy.

DETAILED DESCRIPTION:
This study is intended to carry out a single arm, prospective, open clinical study, and use Darsilide combined with endocrine therapy, Trastuzumab and Patuzumab to treat early or locally advanced breast cancer of TPBC before surgery. It is intended to further explore the efficacy and safety of the new adjuvant treatment for TPBC patients with step-down therapy.

All participants received 150mg of darcilib once a day. Take it continuously for 21 days, then stop taking it for 7 days, with a treatment cycle of 28 days.Letrozole 2.5mg once daily (premenopausal patients treated with OFS).Trastuzumab (8mg/kg first dose, 6mg/kg sequential) and Patuzumab (840mg first dose, 420mg/kg sequential) were administered intravenously every 3 weeks, or fixed-dose combination of pertuzumab and trastuzumab for subcutaneous injection (1200 mg pertuzumab plus 600 mg trastuzumab loading dose in 15 mL, followed by 600 mg pertuzumab plus 600 mg trastuzumab maintenance doses in 10 mL), both administered every 3 weeks, with all patients receiving 8 cycles of treatment. After starting treatment and before surgery, subjects will be monitored through breast MRI to evaluate clinical tumor remission. The primary endpoint was the pCR rate in the group receiving darcilib+letrozole+HP treatment, defined as the proportion of patients who achieved pCR after surgery after neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female initial treatment patients aged ≥ 18 years and ≤ 70 years.
2. ECOG score 0-1 points.
3. Pathologically confirmed as invasive breast cancer, with tumor staging of II-IIIA.
4. HR positive HER-2 positive.
5. The main organs function normally and meet the following standards:

（1）The blood routine examination standards must comply with:ANC ≥1.5×10 9/L；PLT ≥100×109/L；Hb ≥90g/L. （2）Biochemical examination must meet the following standards: TBIL ≤ 1.5 Upper limit of normal value (ULN)；ALT and AST ≤ 1.5 times the upper limit of normal value (ULN)；Alkaline phosphatase ≤ 2.5 times the upper limit of normal value (ULN)；BUN and Cr ≤ 1.5 × ULN and creatinine clearance rate ≥ 50 mL/min； （3）Cardiac ultrasound and echocardiography: Left ventricular ejection fraction (LVEF ≥ 50%).

6. For female patients who have not undergone menopause or surgical sterilization: Agree to abstain or use effective contraceptive methods during the treatment period and at least 7 months after the last administration during the study treatment.

7. Volunteer to join this study and sign an informed consent form.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer.
2. inflammatory breast cancer.
3. Previously received anti-tumor therapy or radiation therapy for any malignant tumor, excluding cured cervical cancer in situ, basal cell carcinoma, or squamous cell carcinoma.
4. Simultaneously receiving anti-tumor therapies in other clinical trials, including endocrine therapy, bisphosphate therapy, or immunotherapy.
5. The patient had undergone major surgical procedures unrelated to breast cancer within 4 weeks before enrollment, or the patient has not fully recovered from such surgical procedures.
6. Individuals who have previously suffered from clinically significant lung diseases, including but not limited to interstitial pneumonia, pneumonia, pulmonary fibrosis, and radiation pneumonia (excluding radiation changes that do not require corrective treatment), or those who have been found to have such diseases through screening period examinations.
7. Serious heart disease or discomfort, including but not limited to the following diseases:

（1）Confirmed history of heart failure or systolic dysfunction (LVEF<50%). （2）High risk uncontrolled arrhythmia（atrial tachycardia，ventricular tachycardia，Higher level atrioventricular block）； （3）Angina pectoris requiring treatment with anti angina drugs； （4）Clinically significant heart valve disease； （5）ECG shows transmural myocardial infarction； （6）Poor control of hypertension (systolic blood pressure>180 mmHg and/or diastolic blood pressure>100 mmHg)； 8. Inability to swallow, intestinal obstruction, or other factors that affect drug administration and absorption.

9. Individuals with a known history of allergies to the drug components of this protocol；Having a history of immunodeficiency, including HIV testing positive, or suffering from other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation.

10. Pregnant and lactating female patients, those with fertility and positive baseline pregnancy test results, or those of childbearing age who are unwilling to take effective contraceptive measures during the entire trial period and within 7 months after the last study medication.

11. Suffering from severe comorbidities or other comorbidities that may interfere with the planned treatment, or any other situation where the researcher deems the patient unsuitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response | Immediately after surgery
  The proportion of patients in this group who achieved pCR after surgery after neoadjuvant therapy

SECONDARY OUTCOMES:
Adverse event occurrence | At the end of one Cycle (each cycle is 28 days)
  The incidence and severity of adverse events (including serious adverse events)
objective response rate | At the end of Cycle 6 (each cycle is 28 days)
  The proportion of patients who achieved CR or PR before surgery after neoadjuvant therapy among all subjects
Residual cancer burden | Immediately after surgery
  Proportion of patients with residual cancer burden score of 0-1 after surgery
Event free survival | 5 years after surgery
  The time interval between enrollment and the first recording of related events, including preoperative disease progression, postoperative disease recurrence, and death from any cause.
Disease free survival | 5 years after surgery
  The time interval between the first day without disease (surgery date) and the first recording of related events, including postoperative disease recurrence and death from any cause.
Distant disease/recurrence free survival | 5 years after surgery
  The time interval between the first day without disease ( surgery date) and the first occurrence of distant recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan cacer hospital, Henan, Henan, China

IPD SHARING:
Plan to Share IPD: No